CLINICAL TRIAL: NCT04545359
Title: Longitudinal Study of the Effects of Neurofeedback Training on the Level of Relaxation in Healthy Population: Characterization at the Electrophysiological and Behavioral Levels
Brief Title: Study on Neurofeedback and Relaxation
Acronym: NEURORELAX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre National de la Recherche Scientifique, France (Other)
Collaborators: Sorbonne University (Other); Institut du Cerveau et de la Moelle Epinière (Unknown); myBrain Technologies (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, Philippe Fossati, University Professor and Hospital Practitioner in psychiatry, Assistance Publique - Hôpitaux de Paris
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: RCB 2017-A02786-47; 17001 (Registry Identifier: CNRS)
Record Dates: First submitted 2020-03-30; First posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Healthy People
Keywords: Neurofeedback; Electroencephalography (EEG); Alpha rhythm; Relaxation; Melomind device; Longitudinal analysis

STUDY DESIGN:
Intervention Model Description: There are two groups : one receives the real neurofeedback task and the second receives a sham neurofeedback.
  This study is double-blind randomized.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All the persons who may interact with the participants and/or implied in the analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurofeedback Group (Experimental): Participants from this group perform actual neurofeedback training, i.e they are instructed to control -- decrease -- in real-time a sound that is inversely related to the amplitude of their own alpha activity, obtained from Melomind EEG signals.
  Interventions: Behavioral: Alpha-based neurofeedback
- Control Group (Sham Comparator): Participants from this group perform sham neurofeedback based on the feedback sounds generated by the participants from the Neurofeedback Group at the same step of the training program.
  Interventions: Behavioral: Sham neurofeedback

INTERVENTIONS:
Behavioral: Alpha-based neurofeedback — Twelve 21-minute sessions (minimum of 1 session and maximum of 3 sessions per week) of auditory alpha-based neurofeedback with the Melomind device developed by myBrain Technologies (France). Recording of felt relaxation, perceived stress level, anxiety level pre-post sessions.
  Electrophysiological: Recording of EEG signals on 32 electrodes every two sessions.
  Arms: Neurofeedback Group
Behavioral: Sham neurofeedback — Twelve 21-minute sessions (minimum of 1 session and maximum of 3 sessions per week) of an auditory sham neurofeedback with the Melomind device developed by myBrain Technologies (France). Sham feedback is based on the real feedback of the participants in the Experimental arm. Recording of felt relaxation, perceived stress level, anxiety level pre-post sessions.
  Electrophysiological: Recording of EEG signals on 32 electrodes every two sessions.
  Arms: Control Group

SUMMARY:
This longitudinal study deals with the characterization of the electrophysiological and behavioral effects of alpha-based neurofeedback training on the brain networks involved in the relaxation process of healthy people.

DETAILED DESCRIPTION:
Despite a growing number of studies dedicated to neurofeedback, the underlying cerebral mechanisms (plasticity phenomena underlying neurofeedback training or learning) are very poorly known. In most of the work on stress and anxiety reduction, the neural parameters on which neurofeedback is performed are low frequency waves like alpha waves. But the effects that an alpha-based neurofeedback has on these waves and more generally on the oscillatory behaviour of the networks involved after the neurofeedback sessions, are very little studied.

Thus, the NEURORELAX study aims to clarify the effects on neurofeedback training at the (electro)physiological level (changes in brain responses in terms of frequency of oscillations, power and location of the cerebral sources of these activities) and/or behavioural level (relaxation and reduced susceptibility to anxiety). It will use the Melomind neurofeedback device as built by myBrain Technologies company, which will make it additionally possible to assess feasibility of neurofeedback training with this reduced mobile device comprising of 2 dry electrodes. For these purposes, the investigators will propose a series of auditory neurofeedback training sessions to the participants, accompanied by electrophysiological (EEG) and clinical measures. The level of relaxation of the subjects will be characterized by self-reported questionnaires and by electrophysiological signal measurement.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary adult subjects, aged 18 to 60
* No known neurological history
* Having an anxiety level higher than 35 on the STAI-YA scale
* Insured under the French social security system
* Signature of the informed consent
* Absence of visual, hearing, sensory or motor deficits incompatible with participation in the study

Exclusion Criteria:

* recreational use of psychotropic drugs
* ongoing anxiolytic / benzodiazepine treatment
* current depressive episode and/or generalized anxiety troubles
* person under guardianship, curatorship or safeguarding of justice or any other measure
* administrative or judicial deprivation of rights or liberty
* pregnant or breastfeeding
* unable to give consent
* person subject to a period of exclusion from further research

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in alpha frequency band power at the end of the 12 neurofeedback training sessions relative to the initial, pre-training, alpha power level. | From the 1st training session until the end of the 12th training session, the time frame of the assessment is 22 days minimum and 96 days maximum, with a minimum of 1 training session and a maximum of 3 training sessions per week.
  Individual EEG power measures in alpha band (between 7 and 13 Hz), performed over several minutes at rest, pre- and post-training, on every session.
Change in alpha frequency band power at post-training relative to pre-training across every training session. | From the 1st training session until the end of the 12th training session, the time frame of the assessment is 22 days minimum and 96 days maximum, with a minimum of 1 training session and a maximum of 3 training sessions per week.
  Individual EEG power measures in alpha band (between 7 and 13 Hz), performed over several minutes at rest, pre- and post-training, on every session.

SECONDARY OUTCOMES:
Change in the EEG power spectrum at the end of the 12 neurofeedback training sessions relative to the initial, pre-training, EEG spectral content. | From the 1st training session until the end of the 12th training session, the time frame of the assessment is 22 days minimum and 96 days maximum, with a minimum of 1 training session and a maximum of 3 training sessions per week.
  EEG signal measurement performed over several minutes at rest, pre- and post-training, on every session; EEG power spectrum analysis between 0.5 and 45 Hz.
Change in the EEG power spectrum at post-training relative to pre-training across every training session. | From the 1st training session until the end of the 12th training session, the time frame of the assessment is 22 days minimum and 96 days maximum, with a minimum of 1 training session and a maximum of 3 training sessions per week.
  EEG signal measurement performed over several minutes at rest, pre- and post-training, on every session; EEG power spectrum analysis between 0.5 and 45 Hz.
Change in anxiety trait after the 12 neurofeedback training sessions relative to before the first training session. | Assessments are performed before the 1st training session (at day 1) and after the 12th training session (at day 22 up to 96, depending on the number of training sessions per week (1 minimum, 3 maximum)).
  Anxiety trait level measured by the State-Trait Anxiety Inventory (Trait evaluation, STAI-YA), before the 1st neurofeedback training session and after the last neurofeedback training session.
Change in affective state after the 12 neurofeedback training sessions relative to before the first training session. | Assessments are performed before the 1st training session (at day 1) and after the 12th training session (at day 22 up to 96, depending on the number of training sessions per week (1 minimum, 3 maximum)).
  Affective state measured by the Positive and Negative Affect Schedule (PANAS), before the 1st neurofeedback training session and after the last neurofeedback training session.
Change in stress level after the 12 neurofeedback training sessions relative to before the first training session. | Assessments are performed before the 1st training session (at day 1) and after the 12th training session (at day 22 up to 96, depending on the number of training sessions per week (1 minimum, 3 maximum)).
  Subjective stress level measured by the Perceived Stress Scale (PSS), before the 1st neurofeedback training session and after the last neurofeedback training session.
Changes in anxiety state at post-training relative to pre-training across every training session. | Assessments are performed before and after every training session; the estimated period of time of assessment is 22 days minimum and 96 days maximum, with a minimum of 1 training session and a maximum of 3 training sessions per week.
  Anxiety state level measured by the State-Trait Anxiety Inventory (State evaluation, STAI-YB) before and after every training session.
Change in relaxation state at post-training relative to pre-training across every training session. | Assessments are performed before and after every training session; the estimated period of time of assessment is 22 days minimum and 96 days maximum, with a minimum of 1 training session and a maximum of 3 training sessions per week.
  Subjective relaxation state measured by a visual analog scale before and after every training session.
Correlation between the changes in electrophysiological measurements and the changes in behavioral measures. | From the 1st training session until the 12th training session (minimum of 22 days and maximum of 96 days, with a minimum of 1 training session and a maximum of 3 training sessions per week).
  Correlation between EEG power spectrum features and scores at behavioral questionnaires and scales, across training sessions.
Changes in EEG power spectrum during the training sessions from the 1st until the 12th sessions. | From the 1st training session until the 12th training session (minimum of 22 days and maximum of 96 days, with a minimum of 1 training session and a maximum of 3 training sessions per week).
  EEG signal measured continuously during the 21 minutes of neurofeedback training, on every session; EEG power spectrum analysis between 0.5 and 45 Hz.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Fossati, Pr, Principal Investigator — Equipe CIA, ICM GH Pitié-Salpêtrière 47 Bd de l'Hôpital 75651 Paris Cedex 13; Nathalie George, Dr, Principal Investigator — CNRS, CENIR MEG-EEG, ICM; Laurent Hugueville, Principal Investigator — CNRS, CENIR MEG-EEG, ICM; Jean-Yves Rotgé, Dr, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Centre de Neuro-Imagerie de recherche (CENIR), ICM, Paris, France

IPD SHARING:
Plan to Share IPD: No